CLINICAL TRIAL: NCT00563914
Title: An Open Label, 4 Escalating Dose, Randomized Multicentre Study Evaluating the Safety and Activity of Ferroquine Associated With Artesunate Versus a Positive Calibrator (Amodiaquine Associated With Artesunate) in African Adult Patients With Uncomplicated Malaria
Brief Title: A Comparative Safety and Activity Study With Ferroquine Associated With Artesunate Versus Amodiaquine Associated With Artesunate in African Adult Patients With Uncomplicated Malaria
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT10420; SSR97193
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Malaria
Keywords: Malaria
MeSH Terms: conditions — Malaria | interventions — ferroquine; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ferroquine (SSR97193)
- 2 (Active Comparator)
  Interventions: Drug: amodiaquine

INTERVENTIONS:
Drug: ferroquine (SSR97193) — associated with artesunate
  Arms: 1
Drug: amodiaquine — associated with artesunate
  Arms: 2

SUMMARY:
The primary objective is to assess the safety of different doses of ferroquine with artesunate (AS) in adult African patients with uncomplicated malaria.

The secondary objectives are to assess activity in reducing parasitemia and the pharmacokinetics of ferroquine and its metabolites.

DETAILED DESCRIPTION:
The study duration is 30 days including a 2 day screening period, a 3 day treatment period with a follow-up period of 25 days. Patients remain hospitalized 4 days.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50 kg and 90 kg with Body Mass Index >18 kg/m²
* Presence of body temperature ≥ 37.5°C or history of fever within the last 24 hours
* Monoinfection with Plasmodium falciparum and parasitemia within the 100 to 200,000/microL

Exclusion Criteria:

* Hypersensitivity to quinoleines or artesunate
* History or presence of any clinically significant disease or symptoms which, in the judgment of the investigator, might confuse the interpretation of the safety and efficacy information
* Splenectomized patients
* Laboratory parameters outside normal ranges
* Presence of HBs antigen, anti-HCV antibodies and anti-HIV 1&2 antibodies
* Cardio vascular and Electrocardiogram parameters outside normal values
* Presence of criteria of complicated malaria
* Permanent vomiting
* Previous treatment within 5 times the elimination half-life of any anti-malaria agents or with any marketed or investigational drugs (including St John's Wort) within 14 days before administration, or within 5 times the elimination half-life of that drug, whichever the longest, especially CYP3A and 2D6 main substrates
* Positive results on urine drug screen for anti-malaria agents (aminoquinolines)
* History of drug or alcohol abuse (alcohol consumption > 40 grams/day ; i. e. 2.5 beers of 33cl with 5 degrees of alcohol)
* Intention to use herbal medicine during the study period
* Immunization injection within last 15 days

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Hepatic safety :ALT, AST, Alkaline Phosphatase, Total Bilirubin | Sreening , baseline, days D3,D5,D6,D7,D9,D14,D21 and D28

SECONDARY OUTCOMES:
Parasite clearance assessed by repeated measurements of parasitemia | Sreening, days D1(T6 and T12),D2 (T0 and T6), D3( T0, T6 and T12) ,D4,D7,D14,D21and D28
Pharmacokinetics of ferroquine assessed by repeated measurement of blood concentration | up to 28 days after last dosing

CONTACTS AND LOCATIONS:
Overall Officials: Christian Supan, MD, Principal Investigator — URM (Unité de Recherches Médicales), Hôpital Albert Schweitzer, BP 118 Lambaréné, Gabon
Locations (2):
- Sanofi-Aventis Administrative Office, Lambaréné, Gabon
- Sanofi-Aventis Administrative Office, Nairobi, Kenya

REFERENCES:
- [Derived] Supan C, Mombo-Ngoma G, Kombila M, Ospina Salazar CL, Held J, Lell B, Cantalloube C, Djeriou E, Ogutu B, Waitumbi J, Otsula N, Apollo D, Polhemus ME, Kremsner PG, Walsh DS. Phase 2a, Open-Label, 4-Escalating-Dose, Randomized Multicenter Study Evaluating the Safety and Activity of Ferroquine (SSR97193) Plus Artesunate, versus Amodiaquine Plus Artesunate, in African Adult Men with Uncomplicated Plasmodium falciparum Malaria. Am J Trop Med Hyg. 2017 Aug;97(2):514-525. doi: 10.4269/ajtmh.16-0731. Epub 2017 Jul 19. PMID 28722611